CLINICAL TRIAL: NCT02448784
Title: Post-marketing Surveillance of Donepezil Hydrochloride - Investigation of Long Term Safety and Efficacy of Aricept as Well as Its Proper Use Information in Patients With Dementia With Lewy Bodies.
Brief Title: Post-marketing Surveillance of Donepezil Hydrochloride - Investigation of Long Term Safety and Efficacy of Aricept as Well as Its Proper Use Information in Patients With Dementia With Lewy Bodies (DLB).
Status: Completed | Type: Observational
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: ART09T
Record Dates: First submitted 2015-05-14; First posted 2015-05-19 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2017-01

CONDITIONS: Dementia With Lewy Body Disease
Keywords: Donepezil Hydrochloride; ARICEPT; Dementia; Lewy bodies; Dementia with Lewy bodies; Post-marketing surveillance
MeSH Terms: conditions — Dementia; Lewy Body Disease | interventions — Donepezil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants with DLB: Participants with DLB who will receive donepezil hydrochloride per approved label.
  Interventions: Drug: Donepezil Hydrochloride

INTERVENTIONS:
Drug: Donepezil Hydrochloride — Initial dose for oral use is 3 mg once daily. The dose is increased to 5 mg after 1-2 weeks. Following at least 4 weeks of dosing at 5 mg, the dose is increased to 10 mg. The dose may be decreased to 5 mg depending on the symptoms of the participant.
  Other Names: Aricept

SUMMARY:
To investigate long term safety (especially about Parkinsonism) and efficacy of donepezil hydrochloride in clinical practice as well as its proper use information in participants with DLB.

ELIGIBILITY:
Inclusion Criteria:

1. Naive participants diagnosed as DLB

Exclusion Criteria:

1. Participants with a history of donepezil hydrochloride product administration in the past
2. Participants who have already been registered in this surveillance
3. Participants with a history of hypersensitivity to any ingredients of donepezil hydrochloride or piperidine derivatives

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Naive participants diagnosed as Dementia with Lewy bodies and administrated Aricept (donepezil hydrochloride)
Sampling Method: Non-Probability Sample
Enrollment: 591 (Actual)
Dates: Start 2015-04-20 (Actual); Primary Completion 2017-03-30 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
Mean Mini-Mental State Examination (MMSE) score | At Week 12
Mean Mini-Mental State Examination (MMSE) score | At Week 24
Mean Mini-Mental State Examination (MMSE) score | At Week 52
Mean Revised Hasegawa's Dementia Scale (HDS-R) score | At Week 12
Mean Revised Hasegawa's Dementia Scale (HDS-R) score | At Week 24
Mean Revised Hasegawa's Dementia Scale (HDS-R) score | At Week 52

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) /adverse drug reactions (ADRs) | From Week 0 to Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Kazuhiro Omata, Study Director — Drug Fostering and Evolution Coordination Department, Corporate Medical Affairs Headquarters, Eisai Co., Ltd.; Syoya Yamakawa, Study Director — Drug Fostering and Evolution Coordination Department, Corporate Medical Affairs Headquarters, Eisai Co., Ltd.
Locations (1):
- Tokyo, Japan